CLINICAL TRIAL: NCT01119534
Title: Comparative Efficacy of the Suppository Composed by Guaiacol, Eucalyptol, Menthol and Camphor Versus Guaiacol Suppository Versus Guaifenesin Syrup in Pediatric Patients With Cough Due the Infectious Origin
Brief Title: Comparative Efficacy of the Suppository Versus Guaiacol Suppository Versus Guaifenesin Syrup in Pediatric Patients With Cough Due the Infectious Origin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Dr. Jose Espin Neto, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-TRN-03(01/10); Version 05 - March 9, 2010
Record Dates: First submitted 2010-04-29; First posted 2010-05-07 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Cough
Keywords: Cough treatment
MeSH Terms: conditions — Cough | interventions — Guaiacol; Eucalyptol; Menthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Transpulmin (Experimental): Suppository composed by guaiacol, eucalyptol, menthol and camphor
  Interventions: Drug: Guaiacol, eucalyptol, menthol and camphor suppository
- Comparator 1 (Active Comparator): Suppository composed by guaiacol
  Interventions: Drug: guaiacol suppository
- Comparator 2 (Active Comparator): Syrup composed by guaifenesin
  Interventions: Drug: Guaifenesin syrup

INTERVENTIONS:
Drug: Guaiacol, eucalyptol, menthol and camphor suppository — 2 times per day
  Arms: Transpulmin
Drug: guaiacol suppository — 2 times per day
  Arms: Comparator 1
Drug: Guaifenesin syrup — 4.19 mL - 4 in 4 hours
  Arms: Comparator 2

SUMMARY:
It is believed that the suppository consisting of guaiacol, menthol, camphor and eucalyptol, by their pharmacological properties already established for each component, has the ability to reduce the signs and symptoms related to upper respiratory infections in a manner equivalent (not inferior) to medicine used as a comparator in this study and higher than the suppository containing only guaiacol concentration of 12.5 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patients that parents or legal guardians agree to their participation in the study and agree on the terms proposed in the IC, signing it;
* Patients aged ≥ (greater than or equal to) 02 years and ≤ (less than or equal to) 6 years, 11 months and 29 days, of any ethnicity, class or social group.
* Patients with acute respiratory disease of upper respiratory viral diseases (URI);
* Patients with productive cough;
* Clinical picture of URI defined by the doctor that started less than 48 hours.

Exclusion Criteria:

* Patients being treated with antibiotics;
* Presence of clinical features of bacterial infection of the upper airways and / or pulmonary (acute bacterial sinusitis, pneumonia, etc.).
* Patients with non-productive cough;
* Treatment with immunosuppressive drugs;
* Presence of any medical condition that, according to the investigator, should prevent the patient from the study;
* Participation in clinical trials in the 12 months preceding the study, according to Resolution 251 (ANVISA), August 7, 1997, item III, sub-item J;
* Patients with serious diseases;
* Patients who require multidrug treatment;
* Presence of other concomitant pulmonary diseases
* History of hypersensitivity to drugs of the same pharmacological classes of substances under investigation;
* Patients with diseases that interfere with lung function, such as cerebral palsy or muscular atrophies;
* Patients under medication or supplement (eg physiotherapy) that may interfere with the cough;
* Patients with severe dysfunction of the hepatorenal function;
* Patients with x-ray of the chest or sinus compatible with picture of bacterial infection;
* Patients with blood cell count suggestive of bacterial infection;
* Changes in laboratory, clinical, physical and / or radiological agents that, judged by investigators, could compromise patient health or reliability of the data.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of cough of infectious origin. | 7 days of treatment.
  During visits (V1, V2, V3 and V4) will be assessed the signs of improvement of cough of infectious origin.

SECONDARY OUTCOMES:
Analysis of parameters for the improvement of infectious cough. | 7 days of treatment.
  During visits (V1, V2, V3 and V4) will be assessed the signs of improvement in difficulty in breathing,quality of sleep,nasal obstruction, food intake and adherence to the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil